CLINICAL TRIAL: NCT06485167
Title: Effect of High-intensity Electromagnetic Energy (HIFEM®), a Non-invasive Treatment of Urinary Incontinence and Pelvic Floor Dysfunction in Women in Primary Care. A Randomized Controlled Study.
Brief Title: Effect of HIFEM® Treatment of Urinary Incontinence in Women in Primary Care. A Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Lena Rindner, PhD, Vastra Gotaland Region
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FOU2023
Record Dates: First submitted 2024-06-19; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Urinary Incontinence; Quality of Life; Menopause; Mental Health Issue; Primary Health Care
Keywords: urinary incontinence; mental health; menopause; sexual health; womens health; primary health care; quality of ife
MeSH Terms: conditions — Urinary Incontinence; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The intervention treatment consists pelvic floor training with high-intensity electromagnetic energy treatment (HIFEM®). HIFEM® is approval and permission of Food and Drug Administration (FDA) and CE of European Union (EU) to treat UI. One HIFEM® treatment includes 12 000 "Kegel exercises" over 28 minutes on an "intervention-chair". The intervention includes six HIFEM® treatments of 28 minutes with one session per week for six weeks. The woman sits fully clothed on the intervention BLT Emsella chair. Before the first treatment, the woman answers questions about the degree of urinary leakage and records the frequency of urinary leakage before treatment and to next treatment.
  Group 1: Active group (AG): Pelvic floor training with electromagnetic energy HIFEM®. Active treatment group (AG): Includes six HIFEM® treatments of 28 minutes at a frequency of one session/week for six consecutive weeks at program level 1 of 2.
Who Masked: Participant
Masking Description: Group 2: Control group (CG): Non-active HIFEM® (sham-treatment) includes six 28-minute treatments with non-active HIFEM®, one treatment/week for a six-week continuous period with setting below therapeutic level (<10% effect). The control group will be placed on the intervention chair in the same way as the active treatment group. The sham treatment will provide some sensation but without active HIFEM technology. The programming for the sham treatment will be amplitude limited, with the setting below the therapeutic level (<10% effect).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental: Group 1 Active Treatment Group (AG) (Active Comparator): Group 1 Active treatment group (AG)
  ● The AG group consists six HIFEM® treatments of 28 minutes at a frequency of one session/week for six consecutive weeks at program level 1 of 2. The woman will be sitting fully clothed on the HIFEM-chair. Before the first treatment, the woman answers questions about the degree of urinary leakage and records the frequency of urinary leakage before treatment and to next treatment.
  Interventions: Device: HIFEM- chair
- Experimental: Group 2 Sham-treatment Control Group (CG) (Sham Comparator): Group 2 Sham-treatment Control Group (CG)
  ● The CG group consists six non-active HIFEM® treatments (sham-treatment) of 28 minutes at a frecquency of one session/week for six consecutive weeks. The sham-treatment will provide some sensation but without active HIFEM technology. The programming for the sham treatment will be amplitude limited, with the setting below the therapeutic level (<10% effect).The participants will be placed on the HIFEM-chair in the same way as the AG group. Before the first treatment, the woman answers questions about the degree of urinary leakage and records the frequency of urinary leakage.
  Interventions: Device: HIFEM- chair

INTERVENTIONS:
Device: HIFEM- chair — The intervention consists of pelvic floor training combined with high-intensity electromagnetic energy treatment (HIFEM®). This includes six HIFEM® treatments (each lasting 28 minutes) with one session per week over six weeks. The woman completes a voiding diary before treatment and one week (±7 days) after treatment. She sits fully clothed on the HIFEM chair.

SUMMARY:
Urinary incontinence (UI) is a condition with involuntary leakage of urine. UI has a significant impact on health related quality of life, poorer sleep quality and sexual function, reduced participation in social and physical activities and is associated with large health care charge. Non-surgical method is always recommended as first action with a step-by-step care starting from non-invasive to more invasive interventions. Systematic overview shows that available non-surgical treatment options in primary care indicated low results in improving effect. HIFEM® technology is a non-invasive method and studies showed significant result on women with UI. For Swedish healthcare HIFEM® is a new medical technology product to treat UI. However, there is a lack of knowledge about the HIFEM® effect in women seeking primary care.

The aim is to evaluate the effect of high-intensity electromagnetic energy (HIFEM®) on pelvic floor muscles, urinary leakage, sexual function, and health-related quality of life in women with urinary leakage in Swedish primary care, as well as to evaluate cost-effectiveness.

The intervention included six 30 minutes HIFEM® sessions once a week over six weeks compared with control group.

The results are expected to lead to effective non-surgical treatment options that can reach many patients, contribute to improving existing routines and can be a new potential way to support health promotion care in primary care and be a cost-effective investment.

DETAILED DESCRIPTION:
Background Urinary incontinence (UI) is a condition with involuntary leakage of urine. UI has a significant impact on health-related quality of life, poorer sleep quality and sexual function, reduced participation in social and physical activities and is associated with large health care charge. Non-invasive method is always recommended as first action with a step-by-step care starting from non-invasive to more invasive interventions. Systematic overview shows that available non-surgical treatment options in primary care indicated low results in improving effect. HIFEM® technology is a non-invasive method and studies showed significant result on women with UI. For Swedish healthcare HIFEM® is a new medical technology product to treat UI. However, there is a lack of knowledge about the HIFEM® effect in women seeking primary care.

Objective:

he aim is to evaluate the effect of high-intensity electromagnetic energy (HIFEM®) on pelvic floor muscles, urinary leakage, sexual function, and health-related quality of life in women with urinary leakage in Swedish primary care, as well as to evaluate cost-effectiveness.

Method:

The study is a randomized controlled trial evaluating the effect of high-intensity electromagnetic energy (HIFEM®) on pelvic floor muscles in women with urinary leakage. The participants are randomized into two groups: a treatment group receiving active HIFEM treatment and a control group receiving non-active treatment (below therapeutic level). The intervention includes six 30-minute HIFEM® sessions, conducted once a week over six weeks, compared to the control group. The study is blinded to the participants.

Expected result:

Implementation of high-intensity electromagnetic energy (HIFEM®) is expected to improve health for women seeking primary care. The results are expected to increase the knowledge of how women's health is affected by short-term care in primary care through increased quality of life, pelvic floor muscle, sexual function and reduce urinary leakage.

The result may improve existing primary care routines for women with urinary incontinence. The results are also expected to lead to effective non-surgical treatment options that can reach many patients, contribute to improving existing routines and can be a new potential way to support health promotion care in primary care and be a cost-effective investment.

ELIGIBILITY:
Inclusion Criteria:

* Woman
* Age 40-70 years
* Any form of UI - stress incontinence (AI), urge incontinence (TI) or mixed urinary incontinence (MUI) according to QUID
* No major language difficulties that prevent understanding and speaking the Swedish language and filling in questionnaires.

Exclusion Criteria:

* Woman with a serious illness such as psychosis, pulmonary insufficiency, epilepsy, severe depression, dementia, is being treated in palliative care, has ongoing drug or alcohol abuse
* Implanted pacemaker or larger metal implant in the body: metal plates, screws, defibrillator and metal implants in the pelvic area or copper coil
* The patient has a piercing between the waist and knees and is not willing to remove it before each treatment
* Pregnant, or planning to become pregnant, at screening or at any time during the study period
* Painful urges
* Bladder emptying difficulties
* Previous malignancy in the abdomen or urinary tract
* Pelvic floor physical therapy, including muscle training and/or electrical stimulation, in a clinical setting within 30 days prior to screening
* Severely overweight (defined as weight > 135 kg)
* Pulmonary insufficiency, defined as difficulty breathing and fatigue, especially during exercise
* Any condition that causes a lack of normal skin sensation in the pelvis, buttocks and lower extremities
* Currently recovering from surgical procedures where muscle contraction may interfere with the healing process
* Currently receiving treatment for a malignant tumor that would interfere with study participation.
* Used the BTL EMSELLA unit before
* The person has urinary incontinence of neurogenic etiology, such as multiple sclerosis, spina bifida, Parkinson's, spinal cord injury, diabetic neuropathy, etc.
* Vaginal prolapse
* Vaginal rejuvenation treatment, including laser treatments and radiofrequency therapy, within 6 months prior to the screening visit

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — If the woman identifies herself as a woman, she fulfills one of the inclusion criteria for participating in the study
Enrollment: 100 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Short time effect of change in health-related quality of life | Change from baseline to one week, three and six months after completed intervention
  Change in health-related quality of life using The Menopause Rating Scale (MRS) and The Short-Form Health Survey (SF-36).
  Validated questionnaires are used measured quality of life:
  MRS: measures occurrence of menopausal symptoms and health-related quality of life. The questionnaire, which consists of 11 questions and brings together menopausal symptoms in total and in three main groups, somatic symptoms, urogenital symptoms and psychological symptoms. The questionnaire indicates severity of symptoms on a 5-point scale. Low prevalence of symptoms indicates 0 points and high prevalence of symptoms 4 points. The total, individual questions and three subgroups are reported.
  SF-36: examines physical and mental health and changes over time. The questionnaire consists of 36 multiple-choice questions that are divided into eight subscales. Points on the subscales are between 0 - 100, higher values indicate better perceived health.
Short time effect of high-intensity electromagnetic energy on pelvic floor muscles and urinary leakage. | Change from baseline to one week, three and six months after completed intervention
  What is the effect of high-intensity electromagnetic energy on pelvic floor musculature and urinary leakage measured by change in score in ICIQ-UI from baseline to one week, three and six months after completed intervention.
  •International Consultation on Incontinence Questionnaire-Urinary Incontinence-Short Form (ICIQ-UI):The ICIQ-UI is a validated form for use to assess female urinary incontinence. The form consists of four questions and calculates a total score from 0 to 21 from three of the four questions. Recommended cut-offs for severity of urinary leakage: mild (1-5), moderate (6-12), severe (13-18) and very severe (19-21). Higher value indicates worse perceived health.
Short time effect of high-intensity electromagnetic energy on pelvic floor muscles and sexual funktion. | Change from baseline to one week, three and six months after completed intervention
  What is the effect of high-intensity electromagnetic energy on pelvic floor musculature and sexual funktion measured by change in score in ICIQ-UI and MRS urogenital symptoms from baseline to one week, three and six months after completed intervention.
  •International Consultation on Incontinence Questionnaire-Urinary Incontinence-Short Form (ICIQ-UI):The ICIQ-UI is a validated form for use to assess female urinary incontinence. The form consists of four questions and calculates a total score from 0 to 21 from three of the four questions. Recommended cut-offs for severity of urinary leakage: mild (1-5), moderate (6-12), severe (13-18) and very severe (19-21). Higher value indicates worse perceived health.
  The ICIQ-UI form is a validated form to assess female patients with urinary incontinence. The MRS assessed urogenital symptoms such as sexual funktion. With this measures, we hope to be able to assess for overall improvement in symptoms after treatment.

SECONDARY OUTCOMES:
Short time effect of high-intensity electromagnetic energy on pelvic floor muscles and social participation | Change from baseline to one week, three and six months after completed intervention
  Change in health-related quality of life using the social participation measured by:
  * The Menopause Rating Scale (MRS): measures occurrence of health-related quality of life. The questionnaire, which consists of 11 questions divided in three main groups, somatic symptoms, urogenital symptoms and psychological symptoms. The questionnaire indicates severity of symptoms on a 5-point scale. Low prevalence of symptoms indicates 0 points and high prevalence of symptoms 4 points.
  * The Short-Form Health Survey (SF-36): examines physical and mental health and changes over time. The questionnaire consists of 36 multiple-choice questions that are divided into eight subscales. Points on the subscales are between 0 - 100, higher values indicate better perceived health.
  * The Hospital Anxiety and Depression Scale (HADS): examines degree of anxiety (HAD-A) and depressive symptoms (HAD-D). The form consists of 14 graded on a 4-point scale. Higher scores indicate higher prevalence of symptoms.
Short time effect of high-intensity electromagnetic energy on physical activity and incontinence | Change from baseline to six months after completed intervention
  Change in health-related quality of life using the physical activity measured by change in score in two forms the MFI-20 and GSLPAQ from baseline to one week, three and six months after completed intervention. With this measures, we hope to be able to assess for overall improvement in symptoms after treatment.
  * Multidimensional Fatigue Inventory-20 (MFI-20). Measures general and mental fatigue (fatigue) with five dimensions of fatigue; general fatigue, physical fatigue, mental fatigue, reduced motivation and reduced activity. The form contains 20 statements on a five-point scale (25).
  * The Godin-Shephard Leisure-Time Physical Activity Questionnaire (GSLPAQ): The patient estimates how many times on average they do strenuous/moderate/light exercise for more than 15 minutes, during a typical 7-day period. The total score is calculated (26).
  With this measures, we hope to be able to assess for overall improvement in symptoms after treatment.
Does mental health improve when treating urinary incontinence with high-intensity electromagnetic energy compared to non-active treatment? | Change from baseline to one week, three and six months after completed intervention
  Change in mental health will be measured with:
  The Stress and Crisis Inventory (SCI-93). Assesses clinical signs of stress both physical and psychological. Assesses symptoms consistent with autonomic dysfunction. Reference values of <25 no dysfunction. Stress level > 25 - autonomic dysfunction - means limitation to varying degrees of ability and resources for normal psychosocial functioning and vocational rehabilitation. At a stress level > 105, the patient has obvious clinical problems as an obstacle to rehabilitation.
  * The Montgomery-Asberg Depression Rating Scale (MADRS-S): examines the degree of depressed mood and depressive symptoms. The questionnaire consists of 9 questions and higher scores indicate higher prevalence of symptoms.
  * The Hospital Anxiety and Depression Scale (HADS): examines degree of anxiety (HAD-A) and depressive symptoms (HAD-D). The form consists of 14 graded on a 4-point scale. Higher scores indicate higher prevalence of symptoms.
Short tile effect on high-intensity electromagnetic energy improve urogenital health and urinary incontinence | Change from baseline to one week, three and six months after completed intervention
  What is the effect of high-intensity electromagnetic energy on urogenital health measured by change in scores in MRS urogential and ICIQ-UI from baseline to one week, three and six months after completed intervention. These questionnaires MRS and ICIQ-UI, provide an overview of symptoms and the severity of discomfort on urogential health and incontinence. With this measures, we hope to be able to assess for overall improvement in symptoms after treatment.
Short time effect on difference regarding incontinence aids after high-intensity electromagnetic energy compared to non-active treatment? | Change from baseline to one week, three and six months after completed intervention
  What is the effect of high-intensity electromagnetic energy on incontinence aids and incontinence from baseline to one week, three and six months after completed intervention. Questionnaire and diary for the assessment of frequency and consumption of incontinence aids.

CONTACTS AND LOCATIONS:
Overall Officials: Lena Rindner, PhD, Principal Investigator — Vastra Gotaland Region

IPD SHARING:
Plan to Share IPD: No
The descriptive data provided will be summary data for each group. The investigators will not show data from single participants.